CLINICAL TRIAL: NCT06864975
Title: Assessing Different FVIII Dose and Frequency in Immune Tolerance Induction (ITI) with ADVATE Among Hemophilia a Boys with Inhibitor (INITIATE Study): a Multicenter Open-label Non-randomized Clinical Trial
Brief Title: Assessing Different FVIII Doses and Frequencies in Immune Tolerance Induction (ITI) with ADVATE Among Hemophilia a Boys with Inhibitor (INITIATE Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Runhui WU (Other)
Responsible Party: Sponsor-Investigator, Runhui WU, Physician in Charge, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITI by ADVATE (INITIATE)
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia a with Inhibitor
Keywords: immune tolerance induction; ADVATE; FVIII inhibitor; hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Low titer inhibitor - Non-daily dose arm (Experimental): Peak inhibitor titer < 5 BU of historical and during ITI treatment Using FVIII (Advate) 50IU/kg.QoD or 100IU/kg.QoD
  Interventions: Drug: Advate®
- Low titer inhibitor - daily dose arm (Experimental): Peak inhibitor titer < 5 BU of historical and during ITI treatment Using FVIII (Advate) 50IU/kg.QD or 100IU/kg.QD
  Interventions: Drug: Advate®
- High titer inhibitor - low dose arm (Experimental): Peak inhibitor titer ≥5BU and <200BU of historical and during ITI treatment Using FVIII (Advate) 50IU/kg.QD or 100IU/kg.QD
  Interventions: Drug: Advate®
- High titer inhibitor - medium or high dose arm (Experimental): Peak inhibitor titer ≥5BU and <200BU of historical and during ITI treatment Usiing FVIII (Advate) ≥ 100IU/kg.QD
  Interventions: Drug: Advate®
- High titer inhibitor with poor prognosis (Experimental): Peak inhibitor ≥200BU of historical and during ITI treatment FVIII (Advate) ≥ 100IU/kg.QD with immunosuppression agent(s)
  Interventions: Drug: Advate®

INTERVENTIONS:
Drug: Advate® — Non-daily dose FVIII 50IU/kg.QoD or 100IU/kg.QoD
  Arms: High titer inhibitor with poor prognosis
Drug: Advate® — Daily dose FVIII 50IU/kg.QD or 100IU/kg.QD
  Arms: High titer inhibitor - low dose arm
Drug: Advate® — Low dose FVIII 50IU/kg.QD or 100IU/kg.QoD
  Arms: High titer inhibitor - medium or high dose arm
Drug: Advate® — Medium and high dose FVIII ≥100IU/kg.QD
  Arms: Low titer inhibitor - Non-daily dose arm
Drug: Advate® — Medium and high dose FVIII ≥100IU/kg.QD with immunosuppressant agent(s)
  Arms: Low titer inhibitor - daily dose arm

SUMMARY:
Hemophilia A is a blood coagulation disorder caused by deficient or dysfunctional clotting factor VIII (FVIII) leading to incomplete haemostasis. Patients with severe Hemophilia A are predisposed to recurrent bleeding episodes (BEs) in joints and soft tissues that culminate in debiltating arthropathy and long-term morbidity. Prophylaxis with plasma-derived or recombinant FVIII concentrates effectively restores FVIII levels in patients with Hemophilia A, and significantly reduces the risk of bleeding. A critical concern for patients receiving FVIII replacement therapy is the development of neutralising antibodies (inhibitors) against the treatment. Inhibitors develop in up to 40% of patients with severe Hemophilia A when first exposed to FVIII treatment, typically within the first 20-30 exposure days (EDs) although a residual risk remains until after 75 EDs. Inhibitors preclude the use of FVIII replacement therapy for prevention and treatment of bleeding.

Eradication of inhibitors therefore remains an important objective for Hemophilia A patients with inhibitors. Immune tolerance induction (ITI) therapy is the only clinically proven strategy for inhibitor eradication, and at least one attempt should be offered to patients with inhibitors. However, while ITI is well-studied and has a 60- 80% success rate, treatment regimens can be expensive and burdensome to patients.

There are limited data on the use of different dose regimen of FVIII ITI in China. The INITIATE Study was designed to observe treatment strategies in patients with hemophilia A with inhibitors, with a focus on evaluating the safety and effectiveness of different dose regimens of ITI. The INITIATE Study includes multiple groups to explore factors that may affect ITI outcomes, and to explore the effects of different treatment methods on patient ITI biomarkers (genomics, transcriptomics, proteins (antibodies).

DETAILED DESCRIPTION:
1. Research Objective and Significance Coagulation factor VIII (FVIII) is a complex multi-domain glycoprotein and a critical cofactor in the pathway intrinsic to the hemostatic system. Hemophilia A (HA) is an X-linked bleeding disorder characterized by a deficiency of functional FVIII due to defects in the F8 gene encoding coagulation protein FVIII. The prevalence of HA in males is approximately 1/5000. About 40% of HA patients are severe (FVIII activity < 0.01 IU/mL). Due to coagulation disorders, these patients may experience spontaneous bleeding or have difficulty in achieving hemostasis after traumatic injuries, and suffer from recurrent bleeding episodes since childhood, thereby leading to joint disabilities, particularly in the knees, elbows, and ankles. In a small number of cases, severe intracranial hemorrhage can occur, which may be fatal [1]. Currently, prophylactic intravenous infusion of exogenous FVIII concentrates, one of the most immunogenic therapeutic proteins, is the gold standard therapy of severe HA [2]. Therefore, after the infusion of therapeutic exogenous FVIII, patients will develop inhibitors, defined as neutralizing antibodies against FVIII, due to the adaptive immune response of the immune system to FVIII antigens. Neutralizing antibodies occur in 25-40% of individuals, and 70% being high-titer inhibitors with serious hazards [3, 4], which lead to the rapid clearance and inactivation of the exogenous FVIII, consequently resulting in the failure of replacement therapy. Hence, patients may experience difficulties in hemostasis, significantly increased treatment cost [5, 6], reduced quality of life, and dramatically increased morbidity and mortality of complications[7, 8]. Although non-factor drugs, such as bispecific antibodies (emicizumab), are not interfered by FVIII inhibitors and can effectively prevent hemorrhage even in the presence of inhibitors, FVIII remains the optimal hemostatic drug either for treatment of severe traumatic hemorrhage or as supportive therapy during surgery. The efficacy of bypassing agents remains uncertain, rFVIIa involves short half-life and high cost, and the combination of aPCC with emercizumab has a risk of thrombotic microangiopathy [9]. Since HA patients may experience severe bleeding and surgical events throughout their lives, the generation of inhibitors remains a major barrier and the most intractable problem in hemophilia treatment. There has been a consensus that patients with inhibitor should undergo a trial of ITI [10]. Inhibitors typically occur within the first 50 exposure days of FVIII replacement therapy [11], particularly the first 20 exposure days [12], and mostly within 6 months to 2 years after FVIII replacement therapy in infancy and childhood. Therefore, the prevention of inhibitor formation and clearance of inhibitors are important issues in the comprehensive management of pediatric hemophilia. A thorough comprehension of the processes underlying inhibitor clearance therapies serve as an essential foundation for the effective prevention and management of inhibitors.
2. Overview of Chinese and International Research Antibodies against FVIII produced in inhibitor-positive hemophilia patients can rapidly bind to exogenous coagulation factor agents and remove or inactivate them. FVIII protein consists of 2332 amino acids, composed of a heavy chain (A1-a1-A2-a2-B domain) and a light chain (A3-a3-C1-C2 domain) through non-covalent linkage. It exists in the peripheral blood circulation in an inactive form, hydrolyzed and cleaved by protease to expose A2, A3 and C1 domains and functional sites. enabling the formation of a complex with activated Factor IX (FIX), which subsequently generates the activated form of FVIII (FVIIIa). The light chain C1 and C2 domains of FVIIIa bind to negatively charged phospholipids on the surface of platelets and/or von Willebrand factor (VWF), creating conditions for hemostatic function [13]. Due to the large molecular structure, unstable conformation and numerous potential antigenic epitopes of FVIII, the antibodies yielded by immune system of hemophilia patients are variable. Current studies have confirmed that inhibitors interfering with coagulation function of FVIII are polyclonal and can target to different domains of FVIII, including A2 domain of the heavy chain and A3, C1 and C2 domains of the light chain [14]. The FVIII epitope targeted by inhibitors may vary among different patients and even at different time points in the same patient [15]. Previous researchers detected the IgG subtypes of FVIII antibodies in the plasma of patients with anti-HA inhibitors by ELISA, and found that the antibody response to FVIII was regardless of subtypes. Among them, IgG4 and IgG1 were the most abundant prominent subtypes. IgG1 was mostly a transient, non-neutralizing and low-titer inhibitor, while IgG4 was mostly a persistent high-affinity high-titer inhibitor [16]. Therefore, FVIII antibodies are conceptually dominated by IgG, with IgG4 being associated with high-titer inhibitors. There are also studies to detect the binding of each Ig subtypes with FVIII by ELISA during inhibitor production process, and it has been known that a small amount of transient IgM and IgA have certain binding ability to FVIII, associated with transient and low-titer inhibitors, suggesting that IgM and IgA also play a role in the inhibitor production process, although the specific role is not clear [17, 18]. Longitudinal tracking of inhibitors has found that in patients with persistent inhibitors, IgG1 antibodies are initially detected, followed by the appearance of IgG3 and then the highest-affinity IgG4 antibodies. Therefore, it is believed that IgG1 antibodies are associated with non-neutralizing or transient FVIII inhibitors, and whether have neutralizing ability is speculated to be related to the binding epitopes of FVIII. Appearance of IgG3 antibodies on the basis of IgG1 antibodies is always associated with high-affinity and persistent IgG4 antibodies against inhibitors [18]. The role of different IgG subtypes in inhibitor clearance remains to be investigated.

Immune tolerance induction (ITI) by frequent intravenous injection of FVIII is the only proven strategy to eliminate inhibitors and restore the hemostatic effect of exogenous FVIII [12]. At present, ITI regimens mainly include three dosing types: high dose (FVIII 200 IU/kg/QD), medium dose (FVIII 100 IU/kg/QD) and low dose (FVIII 50IU/kg/TiW-QoD) [19]. The overall success rate of ITI ranges from 41% to 91% [20-23]. For those inactive to first-line therapy or with extreme high-titer inhibitors, adjuvant immunosuppressant therapy may increase the likelihood of success. Immunosuppressants include anti-CD20 monoclonal antibody (rituximab), steroids, rapamycin and mycophenolate mofetil. Among them, rituximab that depletes B lymphocytes (from pre-B cells to mature B cells) is recommended as the preferred choice upon guidelines.[24] Rituximab in combination with rescue ITI shows an inhibitor eradication rate of 60%-70%.[25-27] Our center has previously proposed a treatment strategy of low-dose ITI combined with rituximab to eradicate high-titer inhibitors of HA (≥5 BU before ITI initiation). It has shown that 35.7% of children received the low-dose ITI regimen alone, and 64.3% of those who showed poor response to ITI received combination therapy with rituximab (ITI-IS regimen). The success rate of patients with single low-dose ITI was 95%, while for those receiving ITI-IS regimen, the success rate after one cycle of rituximab was 52.6%. Therefore, the overall success rate of low-dose ITI combined with a round of rituximab treatment in our site was 67.9% [28]. With follow-up and the development of second-line therapy, particularly multiple cycles of rituximab, we found that ITI success rate was increased to 67.1% after the second cycle of rituximab treatment and 69.7% after the third cycle (unpublished data). Combined with our previous reports, the overall success rate of clearing high-titer inhibitors via low-dose ITI combined with rituximab can be increased to 80%.

For the exploration of FVIII dose and frequency in ITI treatment, an international multicenter, randomized, prospective and controlled study initiated by an ITI registry compared the efficacy and safety of high-dose (FVIII 200 IU/kg.QD) and low-dose (FVIII 50 IU/kg.TiW) regimens in patients with "favorable prognosis". During 3-year follow-up, the success rate of high-dose and low-dose cohorts was approximately 70%. The high-dose group exhibited faster clearance of inhibitor and restoration of normal FVIII pharmacokinetics, while the low-dose group had approximately three times higher bleeding episodes. Therefore, evidence-based ITI data favor high-dose ITI. In our center, medium-dose ITI, as well as medium-dose combined with immunosuppressive agents, is administered.

However, despite the availability of high, medium, and low doses, ITI treatment with FVIII should be continuous. The relationship between the range of FVIII dose and efficacy remains unclear regarding the stratification of difficulty in inhibitor eradication. Clinical outcomes of ITI are influenced by various factors, including age [29], time from inhibitor diagnosis to ITI [22, 30, 31], F8 genotype [32] and inhibitor titers [33-35]. Nevertheless, outcome prediction of ITI remains a complex challenge, and ITI treatment is still imprecise. Although considerable efforts of immune gene polymorphisms [36], HLA types, precise typing of F8 mutations [37] in the risk of inhibitor production has been explored, their role in ITI treatment remain to be investigated. Although the prophylaxis using non-coagulation factors significantly reduces bleeding episodes, the hemostatic ability is restricted as it can only maintain activity relative to FVIII at a "mild hemophilia" level and cannot meet the demands of highly competitive sports, trauma, or major surgery. additionally, the use of non-coagulation factor interfers with conventional inhibitor testing, increasing the difficulty and cost of detection, resulting in low compliance and different follow-up frequencies among children received ITI combination therapy, which is not conducive to the formation of rapid, effective and stable FVIII immune tolerance, preventing the achievement of the goal of restoring FVIII hemostatic ability. Therefore, it is more necessary to identify the risk of patients for ITI treatment under non-coagulation factor therapy , establishing a model for accurate prediction of ITI outcomes and required duration for different-risk patients under different FVIII dosing frequencies, to achieve precise treatment with individualized regimens for inhibitor patients.

There are still about 20% of children with inhibitors cannot be successfully clear inhibitors even when combined with immunosuppressants such as rituximab. Since rituximab mainly depletes peripheral blood B cells (>90%), it has no effect on memory B cells, plasma cells and T cells [38]. Daratumumab, an anti-CD38 human immunoglobulin (Ig) G1κ monoclonal antibody, has shown excellent therapeutic efficacy in multiple myeloma [39]. With unique ability to trigger cytotoxicity and apoptosis of antibody-producing plasma cells, daratumumab has broad-spectrum potential in the treatment of immune-mediated diseases [40]. Among HA inhibitors, rapid clearance of the FVIII inhibitors with daratumumab has been reported [41]. Regarding refractory FVIII inhibitors, with exceptionally high titers (>200 BU or even >1000 BU), the effectiveness, safety, and long-term efficacy of daratumumab still require further investigation.

There is a risk of inhibitor recurrence after successful ITI. According to cohort studies and reports from registry in 2013, the risk of relapse after successful ITI treatment ranges from 0 to 12.5% [42]. The North American Immune Tolerance Registry (NAITR) reported that the recurrence rate of ITI was approximately 15% during a15-years follow-up period [43]. In Grifols ITI study, the recurrence rate was 6.8% during a 9.1-year follow-up [44]. At one-year follow-up of I-ITI, the recurrence rate was 13% [34]. Previous studies in our center showed a recurrence rate of 11.4% after successful ITI, with recurrence occurring when FVIII dose rapidly reduced or prophylaxis was irregular or interrupted, indicating that there is a risk of recurrence with rapidly decreased ITI dose or irregular prophylaxis [28]. The development of non-coagulation factor prophylaxis has led to the discontinuation of FVIII prophylaxis in children with successful ITI treatment. It has reported that some children did have relapse of inhibitors (Capdevilla Haemoph 2021, Doshl Haemoph 2021, Hassan Haemoph 2021). However, there aren't well-established predictors for favorable outcomes regarding inhibitor recurrence after successful ITI, detection of FVIII-specific T cells and B cells may provide relevant suggestions.

In summary, children with HA, current preventive treatments for hemophilia A patients, regardless of the presence of inhibitors, can yield favorable outcomes. Sustaining tolerance to FVIII and achieving hemostasis through FVIII infusion offer long-term benefits. ITI treatment is the only pathway to eradicate inhibitors and achieve FVIII immune tolerance. Currently, ITI treatment remains imprecise. By integrating clinical characteristics of patients, F8 mutations, immune gene polymorphisms, HLA types, identification of patient prognosis for ITI treatment can be achieved. In addition, establishing models for precise prediction of ITI outcomes and the time required for successful inhibitor clearance under different FVIII dose frequencies for patients at different risk levels is of significant theoretical and practical benefits. This study will also explore the eradication method of refractory FVIII inhibitors to provide effective treatment strategies for refractory patients, explore early warning indicators of relapse after successful ITI, and provide prophylaxis suggestions for children at high risk of relapse, to ultimately achieve the goal that all children can have long-term access to effective hemostasis and bleeding prevention via FVIII.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FⅧ:C <2%);
* Positive for FVIII inhibitors;
* No allergic reactions to FVIII concentrates.

Exclusion Criteria:

* Presence of other coagulation-related diseases,
* Hematological disorders,
* autoimmune diseases
* malignancies

Ages: 0 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-21 (Estimated)

PRIMARY OUTCOMES:
Success | within 24 months
  1. Criteria I (Negative FVIII inhibitor): At least two inhibitor titers <0.6 BU/mL;
  2. Criteria II (Normal FVIII Recovery): FVIII recovery rate ≥ 66% of expected;
  3. Criteria III (Normal FVIII Half-Life): FVIII half-life ≥ 6 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's hospitial, Beijing, Beijing Municipality, China